CLINICAL TRIAL: NCT03396679
Title: Can Ultrasound-detected Subclinical Inflammation Explain Patient's Global Assessment of Disease Activity in Psoriatic Arthritis Considered in Remission ?
Brief Title: Disparity Between Ultrasound- and Clinical Findings in Psoriatic Arthritis in Remission
Acronym: PARURE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9855
Record Dates: First submitted 2017-10-13; First posted 2018-01-11 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: PsA Patients Fulfilling CASPAR Criteria in Remission
Keywords: Psoriatic arthritis; remission; ultrasound
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASPAR criteria agreement: PsA patients fulfilling CASPAR criteria in remission as determined by physician with patient and physician's global assessment of disease activity in agreement compare to Ultrasound examination
  Interventions: Other: Ultrasound examination
- CASPAR criteria disagreement: PsA patients fulfilling CASPAR criteria in remission as determined by physician with patient and physician's global assessment of disease activity in disagreement compare to Ultrasound examination
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Evaluation of the Psoriatic Arthritis remission according to patient and physician's global assessment of disease activity are in agreement (CASPAR criteria agreement) or in disagreement (CASPAR criteria disagreement)

SUMMARY:
Comparison of the proportion of Psoriatic arthritis patients in ultrasound remission (i.e. no power Doppler synovitis, tenosynovitis, dactylitis, enthesitis, PD=0) depending on whether patient and physician's global assessment of disease activity are in agreement or in disagreement.

DETAILED DESCRIPTION:
Current data indicate limited correlations between Ultrasound- and clinical findings of inflammation (synovitis, tenosynovitis, dactylitis, enthesitis) in psoriatic arthritis (PsA). This can could be in relation with subjective parameters included in composite clinical scores, such as patient's global assessment of disease activity. Indeed, there is often a disagreement between patient's and evaluator's global assessments of disease activity in psoriatic arthritisPsA. This can reduce the chance to obtain clinical remission, as defined by such composite clinical scores.

Does residual clinical activity assessed by the patient (and not by the evaluator) reflect objective inflammation assessed by ultrasound, or is it in relation with other factors such as fatigue or depression?

Objectives:

Primary end point:

In PsA patients deemed to be in remission according to their assessing consultant rheumatologist (i.e. low physician's global assessment of disease activity), to compare the proportion of patients with persistant persistent ultrasound findings of inflammation (i.e. at least one power Doppler synovitis, tenosynovitis, dactylitis or, enthesitis, "= PD>0") depending on whether patient and physician's global assessments of disease activity are in agreement or in disagreement (disagreement between patient and physician's global assessments defined by a difference on a VAS ≥ 30/100).

Secondary end points :

* Proportion of patients in clinical remission or low disease activity according to different clinical composite scores (DAS28-CRP, SDAI, DAPSA, et MDA) and proportion of patients in ultrasound remission or minimal ultrasound disease activity (defined as a PD-score=0 and a PD-score≤1 respectively), in this population.
* Comparison of rates of clinical remission and ultrasound remission in patients considered or not in remission according to DAPSA criteria
* Correlation between different composite clinical scores (DAS28-CRP, SDAI, DAPSA, MDA) and ultrasound findings (global power Doppler ultrasound sum score combining synovitis, tenosynovitis, enthesitis, then power Doppler ultrasound score for synovitis, tenosynovitis, enthesitis separately) in this population
* Correlation between different Patient Reported Outcomes (PROs such as HAQ, PsAID, DLQI) and ultrasound findings (global power Doppler ultrasound sum score combining synovitis, tenosynovitis, enthesitis, then power Doppler ultrasound score for synovitis, tenosynovitis, enthesitis separately) in this population
* Evaluation of factors associated with ultrasound remission (PD=0) and with minimal ultrasound disease activity (PD≤1)
* Evaluation of factors associated with a disagreement between patient and physician's global assessment of disease activity (patient global assessment on a VAS - physician's global assessment on a VAS ≥ 30/100).

Study design: prospective transversal observational study Inclusion criteria: PsA patients fulfilling CASPAR criteria in remission as determined by physician Exclusion criteria: patient simultaneously included in another study with blinded treatment; Steinbrocker class IV patients Outcome measure : Comparison of the proportion of patients in ultrasound remission (i.e. no power Doppler synovitis, tenosynovitis, dactylitis, enthesitis, PD=0) depending on whether patient and physician's global assessments of disease activity are in agreement or in disagreement

ELIGIBILITY:
Inclusion criteria:

- PsA patients fulfilling CASPAR criteria in remission as determined by physician, with stable treatment

Exclusion criteria:

- patient simultaneously included in another study with blinded treatment; Steinbrocker class IV patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PsA patients fulfilling CASPAR criteria in remission as determined by physician, with stable treatment
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of Psoriasic arthritis remission | 6 months
  In PsA patients deemed to be in remission according to their assessing consultant rheumatologist (i.e. low physician's global assessment of disease activity), to compare the proportion of patients with persistant ultrasound findings of inflammation by Ultrasound examination (i.e. at least one power Doppler synovitis, tenosynovitis, dactylitis, enthesitis, = PD>0) depending on whether patient and physician's global assessments of disease activity are in agreement or in disagreement.

SECONDARY OUTCOMES:
Comparison of proportion of patients in clinical remission to proportion of patients in ultrasound remission (or minimal ultrasound disease activity) | 6 months
  Proportion of patients in clinical remission or low disease activity according to different clinical composite scores (DAS28-CRP, SDAI, DAPSA, et MDA) and proportion of patients in ultrasound remission or minimal ultrasound disease activity (defined as a PD-score=0 and a PD-score≤1 respectively), in this population.
Comparison of clinical remission and ultrasound remission according to DAPSA criteria | 6 months
  Comparison of rates of clinical remission and ultrasound remission in patients considered or not in remission according to DAPSA criteria
Correlation between different composite clinical scores and ultrasound findings | 6 months
  Correlation between different composite clinical scores (Disease Activity Score 28-CRP (DAS28-CRP) in this population
Correlation between different composite clinical scores and ultrasound findings | 6 months
  Correlation of Simplified Disease Activity Index (SDAI ; Score 0 (remission) to 26 (high activity)) in this population
Correlation between different composite clinical scores and ultrasound findings | 6 months
  Correlation of Disease Activity Index for Psoriatic Arthritis (DAPSA ; Score 0 (remission) to 28 (high activity)) in this population
Correlation between different composite clinical scores and ultrasound findings | 6 months
  Correlation of Minimal Disease Activity (MDA ; Score 5/7)) in this population
Correlation between different composite clinical scores and ultrasound findings | 6 months
  Correlation of ultrasound findings (global power Doppler ultrasound sum score combining synovitis, tenosynovitis, enthesitis, then power Doppler ultrasound score for synovitis, tenosynovitis, enthesitis separately) in this population
Correlation between different Patient Reported Outcomes and ultrasound findings | 6 months
  Correlation of PROs such as Health Assessment Questionnaire (HAQ) in this population
Correlation between different Patient Reported Outcomes and ultrasound findings | 6 months
  Correlation of Psoriatic Arthritis Impact of Disease (PsAID) in this population
Correlation between different Patient Reported Outcomes and ultrasound findings | 6 months
  Correlation of Dermatology Life Quality Index (DLQI) in this population
Correlation between different Patient Reported Outcomes and ultrasound findings | 6 months
  Correlation of Pain Catastrophizing Scale (PCS) in this population
Correlation between different Patient Reported Outcomes and ultrasound findings | 6 months
  Correlation of Fibromyalgia Rapid Screening Tool (FIRST) in this population
Correlation between different Patient Reported Outcomes and ultrasound findings | 6 months
  Correlation of ultrasound findings (global power Doppler ultrasound sum score combining synovitis, tenosynovitis, enthesitis, then power Doppler ultrasound score for synovitis, tenosynovitis, enthesitis separately) in this population
Evaluation of factors associated with a disagreement between patient and physician's global assessment of disease activity | 6 months
  Evaluation of factors associated with a disagreement between patient and physician's global assessment of disease activity (patient global assessment on a VAS - physician's global assessment on a VAS ≥ 30/100).

CONTACTS AND LOCATIONS:
Overall Officials: Gaël MOUTERDE, MD, Principal Investigator — Montpellier Hospital
Locations (1):
- CHU Lapeyronie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No